CLINICAL TRIAL: NCT05808699
Title: Camera Qualification of an Additional Fundus Camera Paired With An Autonomous AI for Detecting Diabetic Retinopathy
Brief Title: Camera Qualification Study
Status: Active, not recruiting | Type: Observational
Sponsor: Digital Diagnostics, Inc. (Industry)
Collaborators: Laboratory Corporation of America (Industry)
Responsible Party: Sponsor
Other Study IDs: DXSDR006
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Fundus camera image: Subjects imaged with a fundus camera
  Interventions: Device: handheld fundus camera

INTERVENTIONS:
Device: handheld fundus camera — Fundus camera

SUMMARY:
A multi-center study to evaluate the performance of an automated device for the detection of diabetic retinopathy with the use of an additional fundus camera with IDx-DR.

DETAILED DESCRIPTION:
A multi-center Study to demonstrate non-inferiority of the automated device detecting diabetic retinopathy using a handheld fundus camera with IDx-DR.

ELIGIBILITY:
Inclusion Criteria:

1. 22 years of age or older
2. Documented diagnosis of diabetes mellitus, as per any of the following:

   1. Having met the criteria established by either the World Health Organization (WHO) or the American Diabetes Association (ADA)
   2. Hemoglobin A1c (HbA1c) ≥ 6.5%
   3. Fasting Plasma Glucose (FPG) ≥ 126 mg/dL (7.0 mmol/L)
   4. Oral Glucose Tolerance Test (OGTT) with two-hour plasma glucose (2-hr PG) ≥ 200 mg/dL (11.1 mmol/L), using the equivalent of an oral 75 g anhydrous glucose dose dissolved in water
   5. Symptoms of hyperglycemia or hyperglycemic crisis with a random plasma glucose (RPG) ≥ 200 mg/dL (11.1 mmol/L)
3. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

1. Currently participating in an interventional eye study
2. Has a known allergy to or contraindication for the use of Tropicamide 1% or other mydriatic eye drops
3. Has a condition that, in the opinion of a licensed clinical team member or investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure or glycemic control, microphthalmia or previous enucleation)
4. Pregnancy
5. Self-report of visual symptoms including vision loss or blurred vision that cannot be corrected (e.g., with eyeglasses) or floaters
6. History of laser treatment of the retina, injections into either eye, or any history of retinal surgery
7. Previous confirmed diagnosis of a retinal disease (e.g., macular edema, severe non-proliferative retinopathy, proliferative retinopathy, radiation retinopathy, or retinal vein occlusion)
8. Any condition that is contraindicated for the use of the study camera
9. Contraindication for imaging by devices used in the study due to any of the following:

   1. Subject is hypersensitive to light
   2. Subject recently underwent photodynamic therapy (PDT)
   3. Subject is taking medication that causes photosensitivity

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic - sampling method: non-probability sequential, invitation to volunteer
Sampling Method: Non-Probability Sample
Enrollment: 626 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity Corrected for Enrichment | Day 1
  Estimation sensitivity and specificity corrected for enrichment using logistic regression, Level 1

SECONDARY OUTCOMES:
Observed Sensitivity and Specificity, Level II | Day 1
  Estimation diagnosability, and observed sensitivity and specificity

OTHER OUTCOMES:
Precision substudy | ~1-month after Day 1
  Evaluate the repeatability and reproducibility of IDx-DR with the camera in protocol DXSDR006.
  Additionally, another IRB-approved R&R study (i.e., similar to DXSDR006 precision substudy) was conducted to evaluate parameters that may optimize R&R outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Abramnoff, MD, PhD, Study Chair — Digital Diagnostics, Inc.
Locations (9):
- United States (9):
  - Infinity Clinical Research, Norco, California
  - Dream Team, Pomona, California
  - East Cost Institute for Research, Jacksonville, Florida
  - Ocean Wellness Center, Miami Gardens, Florida
  - Olive Branch Family Medical Center, Olive Branch, Mississippi
  - Logan Health, Kalispell, Montana
  - Lillestol Research, LLC, Fargo, North Dakota
  - Allure Health, Friendswood, Texas
  - Mt. Olympus Medical Research, Sugar Land, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abramoff MD, Lavin PT, Jakubowski JR, Blodi BA, Keeys M, Joyce C, Folk JC. Mitigation of AI adoption bias through an improved autonomous AI system for diabetic retinal disease. NPJ Digit Med. 2024 Dec 19;7(1):369. doi: 10.1038/s41746-024-01389-x. PMID 39702673